CLINICAL TRIAL: NCT05068219
Title: Efficacy of a Contract-Relax Technique in the Physical Therapy Management of Diaphragmatic Paresis After Cardiac Surgery
Brief Title: Contract-Relax (CR) Technique in the Management of Diaphragmatic Paresis After Cardiac Surgery
Acronym: COREDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/01
Record Dates: First submitted 2021-09-24; First posted 2021-10-05 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Surgery, Cardiac
Keywords: Respiratory complications; Diaphragmatic paresis; Contract-Relax technique; Ultrasound measurement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: To minimize assessment bias, investigators and evaluators (doctor and ultrasound operator) will be unaware of the intervention group. Only the physiotherapist, who will realize the procedure, and the patient will know the arm of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual technique (Active Comparator): Standard rehabilitation
  Interventions: Procedure: Usual physical therapy
- CR technique (Experimental): Standard rehabilitation + 3 CR
  Interventions: Procedure: Usual physical therapy; Procedure: Contract-Relax technique

INTERVENTIONS:
Procedure: Usual physical therapy — Standard rehabilitation for diaphragmatic paresis
  * EFA (Expiratory Flow Acceleration) at the upper thoracic level.
  * PEP (Positive Expiratory Pressure).
  * Expectoration if necessary (coughing up and spitting out)
Procedure: Contract-Relax technique — The diaphragmatic CR is done in a semi-sitting position.
  The CR is composed of 4 steps :
  * First maximum inspiration expiration with position of the hands of the physiotherapist on the last ribs and without resistance (Goal: taking rhythm).
  * Second maximum inspiration expiration : Free inspiration, expiration with pressure on the last ribs to bring the diaphragm into internal stroke.
  * Maximum inspiration against resistance, then maximum expiration with increased pressure.
  * Maximum inspiration with dynamic release of resistance (Goal: hyperextension of the diaphragm) followed by maximum expiration with resistance to allow an increase in expiratory flow.
  Arms: CR technique

SUMMARY:
Postoperative respiratory complications are common complications of patients after cardiac surgery and increase morbidity and mortality and hospital length of stay. Diaphragmatic dysfunction accounts for between 2 and 15% of these complications. Diaphragmatic paresis is one of these dysfunctions and could be due to an intra-operative phrenic nerve injury or harvesting of a mammary artery responsible for diaphragmatic devascularization. It alters the ventilatory mechanics and causes acute respiratory distress often requiring the use of mechanical ventilation. The diagnosis of this dysfunction can be made by thoracic ultrasound with assessment of diaphragmatic excursion. For patient with paresis, ultrasound criteria is an excursion < 25 mm after deep inspiration for at least one of the two hemidiaphragms. This dysfunction is most often transient in the postoperative period, but it can also become persistent.

Contract-Relax (CR) physical therapy technique can be applied to any muscle, providing muscle strengthening, neuromotor stimulation, and a gain in joint amplitude.

Currently, post-cardiac surgery management of respiratory physiotherapy is the same for a patient with or without paresis. Moreover, the CR technique of the diaphragm is not part of this "standard" rehabilitation.

The objective of this study is to determine if the CR technique associated with the current respiratory management allows an early rehabilitation of patients with diaphragmatic paresis after cardiac surgery.

DETAILED DESCRIPTION:
This is a single-center, prospective, comparative, randomized, controlled, parallel group, single blind study, trial assessing the efficacy of the association of CR with a "standard" respiratory rehabilitation for patient with diaphragmatic paresis after cardiac surgery.

This study compares two group :

* "Control" group : Standard rehabilitation (4 rehabilitation sessions a day in Intensive Care Unit (ICU) and 2 sessions in cardiac surgery unit).
* "Interventional' group : Standard rehabilitation + 3 CR during each session. A stratification of the randomization is planned according to diaphragmatic involvement (unilateral versus bilateral).

Diaphragmatic excursion will be assessed by thoracic ultrasound in time motion (TM) mode at D3 and D5, before the first physiotherapy session of the day.

The probe is placed on the mid-clavicular line under the costal grill, with an orientation at 90° of the diaphragmatic dome. The aim is to see the diaphragm through an acoustic window: the liver on the right and the spleen on the left. The diaphragm appears as a hyper echogenic line, the excursion is measured with the TM mode.

Oxygen saturation SpO2 will be taken before and after each respiratory physiotherapy session taking place at D3 and D4. A measurement will be taken on D5 before the first rehabilitation session of the day.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery under extracorporeal circulation,
* Postoperative diaphragmatic paresis (Diaphragmatic excursion <25mm),
* Consent for participation,
* Affiliation to the social security system

Exclusion Criteria:

* History of respiratory pathologies,
* History of neurological pathologies,
* Post-operative cardiac and circulatory complications,
* Pregnant or breastfeeding women,
* Unable to understand,
* Guardianship, curators or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic excursion in maximum inspiration | Day 5
  Diaphragmatic excursion ratio in maximum inspiration at D3 and D5. These measurements are determined by ultrasound in TM mode at D3 before the first rehabilitation session of the day (M1max, displacement, mm) and at D5 before the first rehabilitation session of the day (M2max, displacement, mm).

SECONDARY OUTCOMES:
Diaphragmatic excursion in normal inspiration | Day 5
  Diaphragmatic excursion ratio in normal inspiration at D3 and D5. These measurements are determined by TM ultrasound at D3 before the first rehabilitation session of the day (M1rest, displacement, mm) and at D5 before the first rehabilitation session of the day (M2rest, displacement, mm).
Oxygen saturation | Day 5
  SpO2 (%) before and after each physiotherapy session on D3 and D4 and before the first rehabilitation session of the day on D5.
Non-invasive ventilation | Day 30
  Duration of non-invasive ventilation : NIV, optiflow, CPAP (hours).
Oxygenation | Day 30
  Time of oxygen therapy weaning (hours). The reference time t0 will be the time of postoperative extubation.
Incidence of respiratory complications | Day 30
  Occurence of reintubation, lung disease, atelectasis, bronchial fibroscopy, bronchospasm, pleural effusion, pneumothorax.
Intensive care unit ICU length of stay | Day 30
  Duration of ICU stay (days).
Hospital length of stay | Day 30
  Duration of hospitalization (days).
Pain score : Numeric Rating Scale (NRS) | Day 4
  Self-assessment by the patient of the pain felt with a Numeric Rating Scale (NRS) from 0 (No pain) to 10 (Worst Possible Pain) after each session of respiratory physiotherapy at D3 and D4.

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No